CLINICAL TRIAL: NCT02702453
Title: True NTH Sexual Recovery Intervention for Prostate Cancer Survivors and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Emory University (Other); Movember Foundation (Other); Johns Hopkins University (Other); Memorial Sloan Kettering Cancer Center (Other); University of California, Los Angeles (Other); University of North Carolina (Other)
Responsible Party: Principal Investigator, Daniela Wittmann, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00107048
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Sexual Disfunction; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- Development and Testing (Experimental): Develop an online interactive, tailored intervention to address the needs of men and partners interested in sexual recovery after treatment for localized prostate cancer during the first 6 months after treatment. The intervention will undergo content testing through 4 focus groups with prostate cancer survivors and partners and usability testing with 5 survivors and partners
  Interventions: Behavioral: website

INTERVENTIONS:
Behavioral: website — The intervention arm will consist of 12 modules, 8 of which are consistent with the trajectory of prostate cancer and its treatment. Four modules address aspects of the prostate cancer experience that are important for patients and partners as well as providers and are designed to optimize the goal of supporting patients and partners in their sexual recovery.

SUMMARY:
There is increasing evidence that sexual activity is associated with greater resilience and higher well-being in older adults. Even at a time of stress, and even during a late stage of illness, men and their partners turn to sexual intimacy to increase a sense of connection, comfort and support. The Sexual Recovery intervention seeks to address an unmet need of prostate cancer survivors and their partners who are at risk for poor mental health and decreased quality of life as a result of sexual dysfunction.

By using technology, the intervention will be widely accessible to survivors, the majority of whom do not currently have any access to sexual health expertise. The content and format of the intervention seeks to empower prostate cancer survivors and partners with knowledge and strategies to improve their sexual function, sexual confidence and their sexual relationship. The intervention begins prior to and continues following their definitive treatment. This may, in turn, improve mental health and quality of life.

In a broader sense, this intervention will be transferable. With appropriate modifications, it can become an accessible sexual health intervention for populations dealing with other cancers and chronic illnesses.

DETAILED DESCRIPTION:
This proposal is innovative in a number of ways:

* The intervention is based on a full understanding of the complex nature of sexuality with its bio- (functional), psycho- (confidence), and social (relationship components). It incorporates modules that address each of these factors and their inter-dependencies.
* The intervention is sensitive to critical points in sexual recovery and to patient and partner preferences in the context of therapies for prostate cancer. The intervention acknowledges that there are certain time points at which concerns typically arise (e.g., when preparing for definitive treatment). The effectiveness of the intervention is increased by the use of tailoring linked to patient reported outcomes (e.g., decreased erectile function, increases in depression indices) and to patient/partner preferences.
* The intervention includes partners as equal stakeholders in the sexual recovery and legitimizes their needs for sexual fulfillment and support
* The intervention demonstrates a sensitivity to sexual orientation and cultural diversity
* The intervention is scalable and available at limited or no cost to prostate cancer survivors and their partners regardless of geographical location or system of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with localized prostate cancer who are about to receive definitive treatment with either radiation with or without ADT (androgen deprivation therapy) or prostatectomy AND who also have a spouse or been in a committed relationship with their partner for at least 6 months who is willing to participate in the study. Both parties are required to sign an informed consent, able to speak or read English, have reliable internet access,have their own e-mail address, or be willing to sign up for a new one, and must be 18 years of age or older. The participants must be consented at least two weeks prior to the start of treatment, so that participants will have enough time to complete a baseline survey and access the first module of the intervention.

Exclusion Criteria:

* Anyone unable to speak or read English, unwilling to sign an informed consent, under the age of 18, or people without internet access will be excluded from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2016-03; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
PROMIS (Patient-Reported Outcomes Measurement Information System) Sexual Satisfaction | 4 years
  The primary outcome is PROMIS (Patient-Reported Outcomes Measurement Information System) Sexual Satisfaction. Basing power calculation on the average adjusted score (50) and standard deviation (10) provided in the PROMIS scoring, anticipating Sexual Satisfaction scores for the intervention group vs control group to be 50 vs 45, using a two-tailed t-test, power of 80%, and significance level of 0.05, it is expected this study will recruit 128 patients and 128 partners.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Wittmann, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Wittmann D, Mehta A, Northouse L, Dunn R, Braun T, Duby A, An L, Arab L, Bangs R, Bober S, Brandon J, Coward M, Dunn M, Galbraith M, Garcia M, Giblin J, Glode M, Koontz B, Lowe A, Mitchell S, Mulhall J, Nelson C, Paich K, Saigal C, Skolarus T, Stanford J, Walsh T, Pollack CE. TrueNTH sexual recovery study protocol: a multi-institutional collaborative approach to developing and testing a web-based intervention for couples coping with the side-effects of prostate cancer treatment in a randomized controlled trial. BMC Cancer. 2017 Oct 2;17(1):664. doi: 10.1186/s12885-017-3652-3. PMID 28969611